CLINICAL TRIAL: NCT05699785
Title: Comparison of Inflammatory Markers and Incidence of Comorbidities in Patients on Antiretroviral Therapy (ART) With Second-generation Anti-integrase Drugs on Triple Versus Dual Therapy
Brief Title: Comparison of Inflammatory Markers and Incidence of Comorbidities in Patients on Antiretroviral Therapy With Second-generation Anti-integrase Drugs on Triple Versus Dual Therapy
Acronym: COLLATERAL 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-PP-04
Record Dates: First submitted 2022-12-27; First posted 2023-01-26 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — CD4-CD8 Ratio

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients on antiretroviral therapy with second generation anti-integrase drugs in triple therapy (Experimental)
  Interventions: Other: plasma inflammatory markers; Other: CD4/CD8 ratio
- patients on antiretroviral therapy with second generation anti-integrase drugs in dual therapy (Experimental)
  Interventions: Other: plasma inflammatory markers; Other: CD4/CD8 ratio

INTERVENTIONS:
Other: plasma inflammatory markers — Evolution of different plasma inflammatory markers (CRP, IL6, D-Dimers, CD14s, CD163, IL-1, IP-10, MCP-1, IL-18, IFAB)
Other: CD4/CD8 ratio — Evolution of CD4/CD8 ratio

SUMMARY:
HIV-infected patients develop comorbidities earlier than the general population. Immune activation with the secretion of pro-inflammatory cytokines would play a major role in the occurrence of these comorbidities. Numerous factors, called risk factors, already identified in the general population and confirmed in patients with HIV virus favor the occurrence of these comorbidities but cannot alone explain the overrepresentation and precocity of these comorbidities in the HIV population. Investigators hypothesize that optimization or simplification with certain classes of antiretrovirals modify the inflammatory response and are predictive factors for the occurrence of comorbidities

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age > 40 years or adults with more than 10 years of antiretroviral therapy
* Switching to BIC/FTC/TAF or DTG/3TC or DTG+3TC within the last 2 years
* Plasma HIV-1 RNA viral load < 50 copies/ml for more than 6 months
* Absence of chronic hepatitis B infection
* Absence of genotype mutations on Dolutegravir (DTG) or Bictegravir (BIC) or tenofovir alafenamide TAF
* Daily use of antiretroviral therapy
* Effective contraception for women of childbearing potential will be requested
* Signed informed consent
* Enrollment in a Social Security plan

Exclusion Criteria:

* Non-daily or intermittent antiretroviral therapy regimen (e.g., 4 or 5 days a week)
* Pregnancy or breastfeeding
* Vulnerable persons according to article L.1121-6 of the public health code Persons unable to give consent according to article L.1121-8 of the public health code
* Opportunistic infections during curative treatment
* HIV-2 infection
* Active hepatitis C
* Refusal to participate
* Withdrawal of informed consent by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Plasma inflammatory markers | 3 years after baseline
  To measure the evolution of different plasma inflammatory markers (CRP, IL6, D-Dimers, CD14s, CD163, IL-1, IP-10, MCP-1, IL-18, IFAB) over 3 years between the 2 groups.
CD4/CD8 ratio | 3 years after baseline
  To measure the evolution of CD4/CD8 ratio over 3 years between the 2 groups. A CD4/CD8 ratio is considered normal if it is greater than 0.75. Immune hyperactivation occurs when the ratio is below 0.75

SECONDARY OUTCOMES:
Virological failure rate (year 1) | One year after baseline
  Virological failure rate (plasma HIV-1 RNA viral load > 50 copies/ml on two consecutive measurements)
residual viremia rate (year 1) | One year after baseline
  Evolution of the residual viremia rate (detected or quantifiable plasma HIV-1 RNA viral load < 50 copies/ml)
Virological failure rate (year 2) | two years after baseline
  Virological failure rate (plasma HIV-1 RNA viral load > 50 copies/ml on two consecutive measurements)
Residual viremia rate (year 2) | two years after baseline
  Evolution of the residual viremia rate (detected or quantifiable plasma HIV-1 RNA viral load < 50 copies/ml)
Virological failure rate (year 3) | three years after baseline
  Virological failure rate (plasma HIV-1 RNA viral load > 50 copies/ml on two consecutive measurements)
Residuak viremia rate (year 3) | 3 years after baseline
  Evolution of the residual viremia rate (detected or quantifiable plasma HIV-1 RNA viral load < 50 copies/ml)
Prevalence of neuropsychiatric events at 1 year | 1 year after baseline
  To analyze the evolution at 1 year of the prevalence of neuropsychiatric events (including sleep disorders, anxiety, depression) between the two groups from the questionnaires.
Prevalence of neuropsychiatric events at 2 years | 2 years after baseline
  To analyze the evolution at 2 years of the prevalence of neuropsychiatric events (including sleep disorders, anxiety, depression) between the two groups from the questionnaires.
Prevalence of neuropsychiatric events at 3 years | 3 years after baseline
  To analyze the evolution at 2 years of the prevalence of neuropsychiatric events (including sleep disorders, anxiety, depression) between the two groups from the questionnaires.
changes in antiretroviral therapy (year 1) | 1 year after baseline
  Analyze the 1-year change in the prevalence of changes in antiretroviral therapy and the reasons for changes between the two groups based on questionnaires
changes in antiretroviral therapy (year 2) | 2 years after baseline
  Analyze the 2-years change in the prevalence of changes in antiretroviral therapy and the reasons for changes between the two groups based on questionnaires
changes in antiretroviral therapy (year 3) | 3 years after baseline
  Analyze the 3-years change in the prevalence of changes in antiretroviral therapy and the reasons for changes between the two groups based on questionnaires
Evolution of intracellular markers (CD8/CD38, HLA-DR) (year 1) | 1 year after baseline
  To analyze the evolution of intracellular markers (CD8/CD38, HLA-DR) at 1 year between the two cohorts in high-risk subjects (nadir CD4<200 cells/mm3 or history of AIDS stage, or subject aged ≥ 65 years)
plasma markers assay (year 1) | 1 year after baseline
  Analyze the evolution of plasma markers at 1 year between the two cohorts in high-risk subjects (nadir CD4<200 cells/mm3 or history of AIDS stage, or subject aged ≥ 65 years)
plasma markers assay (year 2) | 2 years after baseline
  Analyze the evolution of plasma markers at 2 years between the two cohorts in high-risk subjects (nadir CD4<200 cells/mm3 or history of AIDS stage, or subject aged ≥ 65 years)
plasma markers assay (year 3) | 3 years after baseline
  Analyze the evolution of plasma markers at 3 years between the two cohorts in high-risk subjects (nadir CD4<200 cells/mm3 or history of AIDS stage, or subject aged ≥ 65 years)
risk factors for immune hyper activation | 3 years after baseline
  Analyze and compare risk factors for immune hyper activation (age, CD4 nadir<200 cells/mm3, AIDS stage, residual viremia, archived M184V/I resistance...) in each group
immune activation markers assays and identification of comorbidities | 3 years after baseline
  Correlate immune activation markers with the occurrence of comorbidities
comorbidities (year 1) | 1 year after baseline
  Measurement of the true incidence of major 11 comorbidities (Depression, Cardiovascular, Osteoporosis, Non-AIDS related cancers, Metabolic syndrome, Cognitive disorders, Chronic renal failure , proximal renal tubulopathy, Hepatic fibrosis, Chronic Obstructive Pulmonary Disease, Osteoarthritis) at 1 year
comorbidities (year 2) | 2 years after baseline
  Measurement of the true incidence of major 11 comorbidities (Depression, Cardiovascular, Osteoporosis, Non-AIDS related cancers, Metabolic syndrome, Cognitive disorders, Chronic renal failure , proximal renal tubulopathy, Hepatic fibrosis, Chronic Obstructive Pulmonary Disease, Osteoarthritis) at 2 years
comorbidities (year 3) | 3 years after baseline
  Measurement of the true incidence of major 11 comorbidities (Depression, Cardiovascular, Osteoporosis, Non-AIDS related cancers, Metabolic syndrome, Cognitive disorders, Chronic renal failure , proximal renal tubulopathy, Hepatic fibrosis, Chronic Obstructive Pulmonary Disease, Osteoarthritis) at 3 years
Onset of new comorbidity | 3 years after baseline
  Measure the time to onset of new comorbidity(ies) in each group.
patient profiles | 3 years after baseline
  Describe patient profiles at risk for comorbidities based on different inflammatory biomarkers
individualized and computerized care plan | 3 years after baseline
  Establish an individualized and computerized care plan for the patient after evaluation of the risk factors (according to the profiles) to detect the occurrence or aggravation of comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Durant, Principal Investigator — durant.j@chu-nice.fr
Locations (2):
- France (2):
  - CH Simone VEIL, Cannes
  - CHU Nice, Nice